CLINICAL TRIAL: NCT07038213
Title: Study of Genome-associated Mechanisms of Diabetic Nephropathy and Evaluation of Nephroprotective Therapy in Patients With Type 2 Diabetes Mellitus in the Kazakh Population
Status: Enrolling by invitation | Type: Observational
Sponsor: Astana Medical University (Other)
Collaborators: Viamedis LLP (Unknown)
Responsible Party: Sponsor
Other Study IDs: AP25794125
Record Dates: First submitted 2025-06-09; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus; Diabetic Nephropathy
Keywords: Kidneys; Diabetes; Glycation genes; Kazakhs
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 50 patients with diabetes: 50 patients with diabetes mellitus having kidney disease
  Interventions: Genetic: glycation genes; Diagnostic Test: beta 2 microglobulin
- 50 patients with diabetes mellitus: 50 patients with diabetes mellitus without kidney disease
  Interventions: Genetic: glycation genes; Diagnostic Test: beta 2 microglobulin

INTERVENTIONS:
Genetic: glycation genes — glycation genes
Diagnostic Test: beta 2 microglobulin — b2m

SUMMARY:
The incidence of diabetes remains a serious global health issue, demanding close attention and the development of comprehensive strategies for prevention, early diagnosis, and effective treatment . According to the International Diabetes Federation (IDF), in 2021, the number of people with diabetes reached 537 million, and it is projected to rise to 783 million by 2045. In the Asia-Pacific region, the number of people with diabetes has reached approximately 206 million .

One of the most common complications of diabetes is diabetic nephropathy. In developed countries, such as the United States and European nations, diabetic nephropathy is a leading cause of chronic kidney disease, placing a significant burden on the healthcare system.

In light of this, the development of more effective methods for early detection of diabetic nephropathy remains a relevant objective. Current research focuses extensively on identifying kidney biomarkers that can signal early kidney damage in the disease's initial stages. Moreover, in recent years, genome-wide association studies (GWAS) have shown that diabetic nephropathy has a genetic component and that susceptibility may vary among different ethnic groups. This underscores the need to develop personalized treatments that consider patients' genetic characteristics.

In emerging economies, such as Kazakhstan, the issue of diabetic nephropathy is also becoming increasingly relevant. The rise in diabetes cases, especially in urban populations, has led to a growing number of chronic kidney disease cases and associated disabilities. This results in significant economic costs for the healthcare system, as the treatment of end-stage renal disease patients requires considerable resources. In Kazakhstan, a particularly important aspect is the lack of studies focused on the genetic and clinical characteristics of diabetic nephropathy in the local population.

The project is particularly valuable due to its emphasis on the Kazakh population, which is underrepresented in global studies. This focus allows for the identification of risk factors and specific characteristics of diabetic nephropathy unique to this ethnic group. Such an approach will substantially enhance the country's scientific and technical capacity and boost Kazakhstan's competitiveness on the international scientific stage.

Given the above, research into genome-associated mechanisms of diabetic nephropathy and evaluation of the effectiveness of nephroprotective therapy in patients with type 2 diabetes within the Kazakh population represent scientific novelty and practical significance. Such studies will help improve the effectiveness of therapeutic and rehabilitation measures, contribute to identifying genetic variations specific to the Kazakh population, and improve patients' quality of life. This will also have a positive impact on healthcare economics and enhance patients' quality of life, while contributing to the global genetic data regarding the Kazakh population.

DETAILED DESCRIPTION:
To achieve the goal of the project, the following tasks were formulated, consisting of a subset of direct sequences designed to consistently lead to results. The study of genome-associated mechanisms of diabetic nephropathy and the evaluation of the effectiveness of nephroprotective therapy in patients with type 2 diabetes mellitus in the Kazakh population may provide new diagnostic opportunities and influence treatment options for patients, and this hypothesis has been tested on five proposed tasks:

1. Recruiting research participants.

   * Make a list of potential participants
   * Invitation of respondents of Kazakh nationality
   * Obtaining written informed consent. A preliminary list of project participants will be created together with endocrinologists. The invitation will be carried out by dialing through the list of participants. A written agreement will be received after the participants have familiarized themselves with the progress of the study.
2. Working with respondents.

   * Collecting anamnesis of the disease and life
   * Clinical and diagnostic examination of the study participants. Clinical and diagnostic examinations will be conducted for all participants of the study, as a result of which participants will be selected according to the inclusion and exclusion criteria. As a result, a database of study participants will be created.
3. Conducting a genetic study and a study of the tubular function of the project participants. Glycation genes will be examined from the venous blood samples of the study participants and markers of tubular function such as beta-2 microglobulin, albumin creatinine ratio and Ngal (neutrophil gelatinase-associated lipocalin) will be studied based on urine analysis.
4. The analysis of the results obtained and the study of the effectiveness of nephroprotective therapy in dynamics in the studied patients.
5. Interpretation and publication of the results. Based on the results of this study, articles will be prepared for international peer-reviewed journals (with a non-zero impact factor): at least 2 (two) articles in journals from the first three quartiles by impact factor in the Web of Science database or having a CiteScore percentile in the Scopus database of at least 50.

ELIGIBILITY:
Inclusion Criteria:

* consent of the participant (signing the informed consent form);
* patients with a verified diagnosis of type 2 diabetes mellitus of Kazakh nationality
* age from 18 years to 65 years

Exclusion Criteria:

өage under 18 and over 65 years

* undiagnosed type 2 diabetes mellitus
* lack of informed consent
* pregnancy and lactation at the time of inclusion in the study;
* oncological disease at the time of inclusion in the study, decompensated concomitant somatic pathology.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be consulted by a therapist, an endocrinologist, a nephrologist, a collection of complaints, anamnesis of the disease and life, an objective examination of organs and systems will be carried out.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-19 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
glycation genes | after completion of the study, on average 2 years
  Allele and genotype frequencies

CONTACTS AND LOCATIONS:
Overall Officials: Murzakhmetova Aigerim Orazbayevna Murzakhmetova Aigerim Orazbayevna, PhD, Study Director — Astana Medical University
Locations (1):
- AstanaMU, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT07038213/Prot_SAP_000.pdf